CLINICAL TRIAL: NCT04479189
Title: LAMP Assay Versus PCR for Detection of blaNDM-1 and blaKPC Genes Among Carbapenem Resistant Gram Negative Isolates at Assiut University Hospitals
Brief Title: LAMP Assay Versus PCR for Detection of blaNDM-1 and blaKPC Genes
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ayat Hussein Mohammed, Principal Investigator, Assiut University
Other Study IDs: LAMP Assay
Record Dates: First submitted 2020-07-15; First posted 2020-07-21 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Gene Amplification

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this work is Detection of gram-negative isolates from different clinical samples,determination the antimicrobial susceptibility pattern of gram-negative isolates to various antimicrobial agents, Molecular Detection of blaNDM-1 and blaKPC gene among gram-negative isolates by PCR, Molecular Detection of blaNDM-1 and blaKPC gene among gram-negative isolates by LAMPand,evaluation the use of the LAMP assay for rapid and cost effective detection of the blaNDM-1 and blaKPC gene among gram-negative isolates in comparison with PCR.

DETAILED DESCRIPTION:
Carbapenem resistance in gram-negative bacteria has become a worldwide problem and has caused a global epidemic that continues to grow..

New Delhi metallo-beta-lactamase 1 (NDM-1) enzyme that confers multi-drug resistance is encoded by New Delhi metallo-beta-lactamase 1 gene (blaNDM-1)]. NDM-1inactivates major classes of beta-lactam antibiotics including carbapenems by cleaving b-lactam rings. NDM-1was reported in 11 different bacterial species including Escherichia coli, Klebsiella sp., Shigella boydii and Vibrio cholera indicating the potential of horizontal gene transfer.

Klebsiella pneumoniae carbapenemase (KPC) enzymes, belonging to class A (serine carbapenemases) and inhibited by boronic acid, have rapidly become a global problem among the Enterobacteriaceae, Pseudomonas aeruginosa and Acinetobacter baumannii .

In infectious disease therapy, administration of adequate antimicrobial agents is essential for preventing the emergence and spread of resistant bacteria. However, conventional antimicrobial susceptibility testing (AST), based on bacterial growth, is time consuming; therefore, a rapid, simple assay is needed for the timely selection of appropriate antibiotics in clinical laboratories such as loop-mediated isothermal amplification (LAMP).

LAMP, developed by the Japanese researcher Notomi, is a novel gene amplification method that can complete DNA amplification under isothermal conditions . LAMP is a strand displacement amplification technique , which utilizes a set of 4 to 6 specially designed oligonucleotide primers and a specific DNA polymerase (Bst). Via the process of strand displacement amplification, a dumbbell DNA structure is produced which serves as a template for cycle amplification. The lack of a need for a thermocycler, the speed of the reaction and make LAMP a promising platform for the development of a simple and sensitive near-patient tool for the molecular detection of genes in resource-limited settings.

LAMP is the most popular and well-established nucleic acid amplification technology among alternatives for the polymerase chain reaction (PCR) . The steps of genetic testing include nucleic acid extraction from the specimens, gene amplification, and detection. These steps require considerable skill and expensive equipment and facilities, making convenient testing at any given location difficult. To overcome these limitations, a new gene amplification method, LAMP reaction, was developed which combines rapidity, simplicity, and high specificity .

ELIGIBILITY:
Inclusion Criteria:

* Patients developing signs of infection on or after the third day of hospital admission (Hospital associated infection)

Exclusion Criteria:

* Patients developing signs of infection before the third day of hospital admission (community acquired infection)

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients infected by carbapenem resistant Gram negative bacteria
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-10 (Estimated); Primary Completion 2022-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
evaluate the use of the LAMP assay for rapid and cost effective detection of the blaNDM-1 and blaKPC gene among gram-negative isolates in comparison with PCR | during the procedure
  Molecular Detection of blaNDM-1 and blaKPC gene among gram-negative isolates by PCR and LAMP

CONTACTS AND LOCATIONS:
Overall Officials: Ayat Mohammed, Principal Investigator — Assiut University